

## Consentimento Informado, Esclarecido e Livre para a Investigação Clínica

Considerando a Declaração de Helsínquia da Associação Médica Mundial (Helsínquia 1964, Tóquio 1975, Veneza 1983, Hong Kong 1989, Somerset West 1996, Edimburgo 2000, Seoul 2008 Fortaleza 2013):

| "Impacto da ingestão de uma infusão de funcho pelas mães na cólica infantil em bebés amamentados exclusivamente |
|---|
| com leite materno." |
| Nome do Estudo (em português): |
| Participante/Representante Legal: |
| Nome: |
| BI/CC n.°: |
| Recebi folheto informativo, tendo ficado ciente dos seus objetivos e do método que irá ser utilizado. |
| Compreendi os riscos que o estudo pode envolver e quais os benefícios que poderão vir a ser alcançados com o mesmo. |
| Tive oportunidade para esclarecer dúvidas, permitindo ter uma decisão mais consciente. |
| Fui informado da possibilidade de livremente recusar ou abandonar a todo o tempo a participação no estudo, sem que |
| isso possa ter como efeito qualquer prejuízo na assistência que me é prestada. |
| Aceito participar neste estudo, de acordo com os esclarecimentos que me foram prestados, tendo recebido uma cópia deste documento. |
| dotto documento. |
| Angra do Heroísmo/Praia da Vitória |
| de de |
| (Assinatura) |
| Investigador: |
| Nome: |
| BI/CC n.º: |
| Confirmo que expliquei ao participante/representante legal, de forma adequada e compreensível, a investigação |
| referida acima, os benefícios, os riscos e as possíveis complicações associadas à realização do mesmo. |
| Informação escrita, em anexo: □ Não □ Sim (n.º de páginas: ) |
| Angra do Heroísmo/Praia da Vitória |
| de de |
| (Applies town) |
| (Assinatura) |